CLINICAL TRIAL: NCT06337916
Title: The Effect of Cervical Stabilization Exercises on the Sense of Cervical Proprioception in Patients With Chronic Neck Pain
Brief Title: The Effect of Cervical Stabilization Exercises on the Cervical Proprioception in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şenay Özdolap (Other)
Collaborators: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Sponsor-Investigator, Şenay Özdolap, Clinical Professor, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/16-01
Record Dates: First submitted 2022-11-07; First posted 2024-03-29 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain; Chronic Neck Pain
Keywords: Chronic Neck Pain; Cervical Stabilization Exercises; Cervical Proprioception
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Stabilization Exercise Group (Active Comparator): 1. The patients age is between the ages of 18-55
  2. Being literate and with good cognitive function,
  3. Having neck pain longer than 3 months
  4. Not taking painkillers and nsaid in the last 1 week
  Interventions: Behavioral: Cervical Stabilization Exercise
- Cervical Standard Exercise Group (Active Comparator): 1. The patients age is between the ages of 18-55
  2. Being literate and with good cognitive function,
  3. Having neck pain longer than 3 months
  4. Not taking painkillers and nsaid in the last 1 week
  Interventions: Behavioral: Cervical Standard Exercise Group

INTERVENTIONS:
Behavioral: Cervical Stabilization Exercise — The cervical stabilization exercise group will receive cervical stabilization exercises 1 session a day, 3 days a week for 6 weeks. Patients will do their exercises in the first 3 weeks accompanied by a physiotherapist, and in the last 3 weeks as a home exercise program.Before the start of the treatment, at the end of the 3rd week and at the end of the 6th week; pain intensity, level of neck disability, quality of life, cervical range of motion and cervical joint position sense will be evaluated and both groups will be compared in these parameters.Demographic information of the patients to be included in the study will be recorded . The patients will be compared to evaluate for Visual Analogue Scale (VAS), Neck Disability Index (NDI) and Short Form (SF-36), cervical range of motion and cervical joint position sense after intervention. Cervical range of motion and cervical joint position sense will be evaluated with the Cervical Range of Motion Deluxe Device (CROM).
  Arms: Cervical Stabilization Exercise Group
Behavioral: Cervical Standard Exercise Group — The patients in cervical standard exercise group will receive conventional cervical exercise for 6 weeks, 3 days a week, 1 session a day. Patients will do their exercises in the first 3 weeks accompanied by a physiotherapist, and in the last 3 weeks as a home exercise program.Before the start of the treatment, at the end of the 3rd week and at the end of the 6th week; pain intensity, level of neck disability, quality of life, cervical range of motion and cervical joint position sense will be evaluated and both groups will be compared in these parameters.Demographic information of the patients to be included in the study will be recorded . The patients will be compared to evaluate for Visual Analogue Scale (VAS), Neck Disability Index (NDI) and Short Form (SF-36), cervical range of motion and cervical joint position sense after intervention. Cervical range of motion and cervical joint position sense will be evaluated with the Cervical Range of Motion Deluxe Device (CROM).
  Arms: Cervical Standard Exercise Group

SUMMARY:
Neck pain is one of the most common musculoskeletal complaints and its prevalence is between 10-22%. Approximately half of all individuals will experience a clinically important neck pain episode over the course of their lifetime. Neck pain is categorized by duration as acute, subacute and chronic neck pain (acute, <6 weeks; subacute, ≤3 months; chronic, >3 months). Chronic neck pain is more common in women and its incidence increases with age. Cervical disc herniation, cervical spondylosis, cervical stenosis, myofascial pain syndrome, cervical instability, whiplash injury, Klippel feil syndrome, thoracic outlet syndrome, cervical sprain, cervical strain, tumors, rheumatic diseases, torticollis, inflammatory neck pain are the main causes.

Anterior tilt of the head is a common posture in neck pain. In this posture, the upper cervical vertebrae are extension, the lower cervical vertebrae are flexion and the cervical lordosis is decreased. With neck pain, inhibition occurs in the deep neck flexor (longus coli and capitis) and extensor (multifidus, rotator, semispinalis) muscles, increased fat infiltration, deterioration in type 1 and 2 fiber ratios, and muscle atrophy. The risk of micro and macro trauma increases and muscle support decreases. Thus, there is an increase in the activation response and fatigue of the neck superficial muscle group (trapeze, scalene, sternocleidomastoid muscles), and a decrease in neck joint movement and proprioception sense. As a result, it was determined that there are deficiencies in the sense of proprioception in patients with neck pain.

Studies have shown that many receptors related to the sense of position are on deep cervical flexor muscles such as Musculus Longus Capitis and Musculus Longus Colli. In cases where there are changes such as atrophy and fat infiltration in these muscles, there is a decrease in proprioceptive sensation.Conservative treatment is the first choice in the treatment of neck pain. The important components of this treatment are stretching, strengthening, posture, stabilization, proprioception, relaxation, joint movement exercises and aerobic exercises. The purpose of stabilization exercises, which have been used in the treatment of chronic neck pain recently; to support the vertebral column by activating the stabilizing muscles and to improve posture by increasing kinesthetic awareness.

This study will examine the relationship between the sense of cervical proprioception and cervical stabilization exercises in patients with chronic neck pain.

In this study, between 15 June 2022 and 30 January 2023; 72 volunteers, aged between 18-55 years, with neck pain for more than 3 months, with good cognitive function, who applied to the our Physical Medicine and Rehabilitation Clinic will be included. The patients will be randomized to two groups as cervical stabilization exercise group and conventional cervical exercise treatment group. The patients in group 1 will receive cervical stabilization exercises 1 session a day, 3 days a week for 6 weeks, and the patients in group 2 will perform cervical stabilization exercises for 6 weeks, 3 days a week, 1 session a day. conventional cervical exercises will be given. Patients of both groups will do their exercises in the first 3 weeks accompanied by a physiotherapist, and in the last 3 weeks as a home exercise program.

Before the start of the treatment, at the end of the 3rd week and at the end of the 6th week; pain intensity, level of neck disability, quality of life, cervical range of motion and cervical joint position sense will be evaluated and both groups will be compared in these parameters.

Demographic information (address, telephone, age, occupation, height, weight, marital status, etc.) of the patients to be included in the study will be recorded and general musculoskeletal examinations will be performed. The patients will be compared to evaluate for Visual Analogue Scale (VAS), Neck Disability Index (NDI) and Short Form-36 (SF-36), cervical range of motion and cervical joint position sense after intervention. Cervical range of motion and cervical joint position sense will be evaluated with the Cervical Range of Motion Deluxe Device (CROM).

ELIGIBILITY:
Inclusion Criteria:

1. The patients age is between the ages of 18-55
2. Being literate and with good cognitive function,
3. Having neck pain longer than 3 months
4. Not taking painkillers and nsaid in the last 1 week

Exclusion Criteria:

1. Cervical extruded or sequestered disc herniation, diagnosis of myelopathy
2. Having neck and shoulder surgery
3. Diagnosis of major trauma, infection, malignancy, inflammatory disease or peripheral nerve compression, spinal congenital anatomical deformity
4. Having severe cardiovascular disease, neurological or mental illness and inability to tolerate treatment
5. Kyphoscoliosis
6. Osteoporosis
7. Stage 3-4 osteoarthritis
8. Diagnosis of diabetes mellitus, uncontrolled hypertension
9. Having a diagnosis of fibromyalgia
10. Spinal stenosis
11. Pregnancy
12. Receiving physical therapy in less than 3 months
13. Obesity (BMI>30)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
assessment of cervical joint position sense | 6 weeks
  Cervical joint position sense will be evaluated with the CROM (Cervical Range of Motion) Deluxe Device.

SECONDARY OUTCOMES:
assessment of cervical range of motion | 6 weeks
  Cervical range of motion will be evaluated with the CROM (Cervical Range of Motion) Deluxe Device.
assessment of neck disability | 6 weeks
  The patients will be evaluate with the Neck Disability Index (NDI) for assessment of neck disability. The score ranges from 0 to 50. As the score increases, disability increases.
assessment of pain | 6 weeks
  The patients will be evaluate with the Visual Analogue Scale (VAS) for assessment of pain. They are numbered from 1 to 10. As the score increases, pain intensity increases.
assessment of life quality | 6 weeks
  The patients will be evaluate with the Short Form (SF-36) for life quality. The SF-36 consists of 36 items - that are grouped in 8 subscales or domains: Physical functioning (10 items); Role limitations due to physical health (4 items); Role limitations due to emotional problems (4 items); Energy/fatigue (4 items); Emotional well-being (5 items); Social functioning (2 items); Pain (2 items); General health (5 items). Scoring is between 0-100, higher scores indicate good health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)